CLINICAL TRIAL: NCT06014983
Title: Efficacy and Adverse Side Effects of Two Forms of Iron in Prenatal Micronutrient Supplements (EASE-Iron): A Randomized Controlled Trial
Brief Title: Efficacy and Adverse Side Effects of Two Forms of Iron in Pregnancy
Acronym: EASE-Iron
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Crystal Karakochuk, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H23-00016
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; Iron Deficiency
Keywords: Iron; Pregnancy; Nutrition
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous fumarate; ferrous bisglycinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous fumarate (Active Comparator): 24 mg elemental iron/day
  Interventions: Dietary Supplement: Ferrous fumarate
- Ferrous bisglycinate (Experimental): 24 mg elemental iron/day
  Interventions: Dietary Supplement: Ferrous bisglycinate

INTERVENTIONS:
Dietary Supplement: Ferrous fumarate — Participants will supplement with 24 mg elemental iron in the form of ferrous fumarate daily for a minimum of 12 weeks.
  Arms: Ferrous fumarate
Dietary Supplement: Ferrous bisglycinate — Participants will supplement with 24 mg elemental iron in the form of ferrous bisglycinate daily for a minimum of 12 weeks.
  Arms: Ferrous bisglycinate

SUMMARY:
This two-arm, double-blind randomized clinical trial will recruit 172 generally healthy, low-risk pregnant individuals aged 19-42 years living in Vancouver, Canada. Participants will be randomized to receive one of two forms of iron (ferrous fumarate or ferrous bisglycinate) in addition to a prenatal multivitamin (without iron) daily during their pregnancy until delivery, with optional continuation until ~4 weeks postpartum for breastmilk sample collection. Blood samples will be taken at baseline (13-25 weeks gestation) and follow-up (35-37 weeks gestation) to assess how different forms of iron impact body iron stores. Stool samples will be obtained within 1 week of both baseline and follow-up visits to assess changes in gut microbiome composition. This research will inform more specific guidelines for optimal iron supplementation practices for the prevention and treatment of iron deficiency for both mother and baby.

DETAILED DESCRIPTION:
To address our primary aim of determining the optimal form of iron in prenatal supplements, we seek to answer the following research questions:

1. Does providing a more bioavailable form of iron (24 mg elemental iron as ferrous bisglycinate) effectively increase ferritin concentration in maternal venous blood and umbilical cord blood, as compared to the standard 24 mg elemental iron as ferrous fumarate?
2. Does 12 weeks of 24 mg daily oral iron as ferrous fumarate increase biomarkers of potential harm (adverse side effects, gut microbiome composition, gut inflammation) in pregnant individuals, as compared to 24 mg daily oral iron as ferrous bisglycinate?

Pregnant individuals 13-25 weeks gestation will be randomized to one of two trial arms to receive either 24 mg elemental iron as ferrous fumarate or 24 mg elemental iron as ferrous bisglycinate for a minimum of 12 weeks during pregnancy until delivery, with optional continuation until 4-weeks postpartum for breastmilk collection. All participants will also receive the standard form and dose of other critical micronutrients during pregnancy (e.g., folic acid, calcium) through the provision of a prenatal multivitamin (not containing iron).

Interested individuals may undergo the informed consent process anytime prior to 25 weeks gestation. Once an individual indicates that they are interested in participating in the trial, the individual will be assigned a unique study ID and a baseline visit will be scheduled.

The baseline visit will occur between 13-25 weeks gestation and will involve discontinuation of current iron/prenatal vitamin supplementation, review and signing the informed consent form (a scanned copy will be shared with the participant), randomization to an iron group, provision of study supplements, completion of a baseline questionnaire, measurement of weight and height, a small blood draw, and provision of a stool collection kit for at-home stool collection.

The intervention period is a minimum of 12 weeks (from baseline at 13-25 weeks to delivery). Participants will supplement daily with the iron and prenatal multivitamin supplements. Monthly follow-up surveys will be sent to participants via email to check-in and receive updates regarding any changes to medical history or medication use.

The follow-up visit will occur between 35-37 weeks gestation and will involve collecting any remaining supplements (for capsule counts and assessment of adherence), a weight measurement, a small blood draw, provision of at-home stool collection kit, and completion of a short follow-up questionnaire.

Optional continuation of study: After the follow-up visit, participants who are planning to breastfeed will have the option to continue supplementing with the study supplements and provide a prenatal colostrum sample and/or 4-week postpartum breastmilk sample.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individual (singleton pregnancy)
* 19-42 years of age
* Living in the greater Vancouver area and willing to travel to the University of British Columbia or BC Women's Hospital for study visits
* 13-25 weeks gestation
* Willing to participate and able to provide informed consent

Exclusion Criteria:

* Having a pre-existing medical condition known to impact iron status (e.g., inherited hemoglobin disorder (i.e., sickle cell, hemochromatosis, thalassemia or other structural hemoglobin variant), malabsorptive disorders (i.e., chronic pancreatitis, cystic fibrosis, celiac disease) and inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis), gastric bypass surgery, atrophic gastritis, advanced liver disease, kidney dialysis)
* Using medications known to interfere with iron metabolism or the gut pathogen equilibrium (e.g., chronic use of proton pump inhibitors, anti-inflammatory agents, non-steroidal anti-inflammatory drugs, antibiotics)
* Having a personal neural tube defect (NTD) history or a previous NTD pregnancy
* Receiving ongoing blood transfusions
* Currently smoking or having smoked in the past 3 months
* Pre-pregnancy body mass index (BMI) ≥30 kg/m^2
* Allergy to any study supplement ingredients

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Maternal ferritin concentration | Blood sample collected at baseline (13-25 weeks gestation) and at follow-up (35-37 weeks gestation)
  µg/L; reflects body iron stores

SECONDARY OUTCOMES:
Maternal hemoglobin concentration | Maternal blood sample collected at baseline (13-25 weeks gestation) and at follow-up (35-37 weeks gestation)
  g/L; obtained through a complete blood count
Umbilical cord ferritin concentration | Umbilical cord blood collected at time of delivery
  µg/L; proxy measure for newborn iron stores
Umbilical cord hemoglobin concentration | Umbilical cord blood collected at time of delivery
  g/L; measured using a HemoCue device
Placental iron concentration | Placenta collected at time of delivery
  µg/g; reflects iron transfer to fetus
Gut microbial analysis | Stool sample collected at baseline (13-25 weeks gestation) and at follow-up (35-37 weeks gestation)
  16S rRNA gene sequencing and targeted real-time PCR (qPCR); gut microbiome composition
Adverse side effects | Follow-up (35-37 weeks gestation)
  Includes reported gastrointestinal side effects (e.g., constipation, diarrhea, nausea) and any other side effects experienced
Markers of inflammation | Maternal blood sample collected at baseline (13-25 weeks gestation) and at follow-up (35-37 weeks gestation); umbilical cord blood sample collected at time of delivery
  Includes alpha-1 acid glycoprotein (AGP; g/L) and C-reactive protein (CRP; mg/L), used in combination to adjust ferritin concentration
Hepcidin concentration | Maternal blood sample collected at baseline (13-25 weeks gestation) and at follow-up (35-37 weeks gestation); umbilical cord blood sample collected at time of delivery
  nmol/L; hormone that influences iron regulation
Breastmilk iron stores | Breastmilk sample collected at 4-weeks postpartum
  Includes measurement of breastmilk iron content (mg/mL) and lactoferrin (mg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Karakochuk, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - BC Women's Hospital, Vancouver, British Columbia
  - University of British Columbia, Food, Nutrition and Health Building, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request, the Principal Investigator will share de-identified individual participant data.